CLINICAL TRIAL: NCT02017899
Title: A Phase 1, Randomized, Observer Blinded, Placebo Controlled, Single Center, Dose Escalation Study to Evaluate the Safety and Immunogenicity of 3 Vaccinations With Shigella Sonnei Vaccine (1790GAHB) Administered Intramuscularly in Healthy Adults.
Brief Title: A Phase 1, Dose Escalation Study, to Evaluate a New Shigella Sonnei Vaccine in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GSK Vaccines Institute For Global Health S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H03_01TP
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-08

CONDITIONS: Shigellosis
Keywords: prevention; Shigella sonnei
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- S. sonnei 1790GAHB - 1 mcg (Experimental): Subjects enrolled in COHORT A receiving 3 injections of S. sonnei 1790GAHB - 1 mcg
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 5 mcg (Experimental): Subjects enrolled in COHORT B receiving 3 injections of S. sonnei 1790GAHB - 5 mcg
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 25 mcg (Experimental): Subjects enrolled in COHORT C receiving 3 injections of S. sonnei 1790GAHB - 25 mcg
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 50 mcg (Experimental): Subjects enrolled in COHORT D receiving 3 injections of S. sonnei 1790GAHB - 50 mcg
  Interventions: Biological: S. sonnei 1790GAHB
- S. sonnei 1790GAHB - 100 mcg (Experimental): Subjects enrolled in COHORT E receiving 3 injections of S. sonnei 1790GAHB - 100 mcg
  Interventions: Biological: S. sonnei 1790GAHB
- Placebo (Placebo Comparator): 2 subjects enrolled in each COHORT A, B, C, D, E receiving 3 injections of Placebo. These were pooled in one Placebo group in the analyses
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: S. sonnei 1790GAHB
  Other Names: Shigella sonnei vaccine
  Arms: S. sonnei 1790GAHB - 1 mcg; S. sonnei 1790GAHB - 100 mcg; S. sonnei 1790GAHB - 25 mcg; S. sonnei 1790GAHB - 5 mcg; S. sonnei 1790GAHB - 50 mcg
Biological: Placebo
  Arms: Placebo

SUMMARY:
This Phase 1 clinical trial is aimed to evaluate the safety and immunogenicity of 3 doses of 5 sequentially escalating dosages of a candidate vaccine against Shigella sonnei (1790GAHB vaccine) administered by intramuscular route in healthy adults (18 to 45 years of age at enrollment). The safety profile of the 1790GAHB vaccine is evaluated in comparison to that of placebo (GAHB-Placebo), constituted by an aluminum hydroxide suspension having the same concentration as study vaccine formulations. A total of 50 eligible subjects will be assigned to one of five sequential cohorts of 10 subjects each.

Within each cohort, in an observer-blind fashion, subjects will be randomized to receive three vaccinations, four weeks apart, of either 1790GAHB vaccine (at five antigen concentrations) or GAHB placebo. A Data Safety Monitoring Board will be in place to receive a summary of all safety data obtained during one week follow-up post-first vaccination with the lower dose. Based on evaluation of the safety data, the Data Safety Monitoring Board will make a recommendation, as to whether the next cohort should be vaccinated with higher antigen concentration or not.

Expected duration of the study for an individual subject is 9 months. Each subject will be followed-up for 6 months after the 3rd vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of age ≥18 years to ≤45 years.
2. Individuals who, after the nature of the study has been explained to them, and prior to any protocol specific procedures being performed, have given written consent according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of medical history, physical examination, hematological / hematochemical blood tests (including presence of high antibody titers against S. sonnei by agglutination test), urinalysis and clinical judgment of the investigator.
4. If women of child-bearing potential, have a negative pregnancy test prior study vaccination and willingness to use acceptable birth control measures for the entire study duration.
5. Individuals affiliated to a social security regimen.

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
2. Individuals with any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
3. Individuals who are not able to understand and to follow all required study procedures for the whole period of the study.
4. Individuals with history of any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
5. Individuals human leukocyte antigen (HLA) -B27 positive and/or with history of reactive arthritis.
6. Individuals with known or suspected HIV infection or HIV related disease, with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system, or under immunosuppressive therapy including use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids (i.e. prednisone, or equivalent ≥10 mg/day) within the previous 28 days, or in chemotherapy treatment within the past 168 days.
7. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
8. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
9. Individuals who have any malignancy or lymphoproliferative disorder.
10. Individuals with history of allergy to vaccine components.
11. Individuals participating in any clinical trial with another investigational product 28 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
12. Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within the entire study duration except influenza vaccination, which is not allowed within the period included between 28 days before 1st vaccination and 28 days after 3rd vaccination.
13. Individuals who have received blood, blood products, and/or plasma derivatives including parenteral immunoglobulin preparations in the past 12 weeks.
14. Individuals who are part of study personnel or close family members to the personnel conducting this study or employees of the clinical trial site institution.
15. Individuals with body temperature > 38.0 degrees Celsius within 3 days of intended study vaccination.
16. Individuals with Body Mass Index (BMI)> 30 kg/m2
17. Individuals with history of substance or alcohol abuse within the past 2 years.
18. Women who are pregnant or are breast-feeding, or are of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study.
19. Females with history of stillbirth, neonatal loss, or previous infant with anomaly.
20. Individuals who have a previously laboratory confirmed or suspected disease caused by S. sonnei.
21. Individuals who have had household contact with/and or intimate exposure to an individual with laboratory confirmed S. sonnei.
22. Any condition, which, in the opinion of the investigator may pose an increased and unreasonable safety risk to the subject if participating to the present study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Prof, Principal Investigator — Centre d'Investigation Clinique en Vaccinologie Cochin-Pasteur (CIC1417)
Locations (1):
- Centre d'Investigation Clinique en Vaccinologie Cochin-Pasteur (CIC1417), Paris, Paris Cedex 14, France

REFERENCES:
- [Derived] Micoli F, Rossi O, Conti V, Launay O, Scire AS, Aruta MG, Nakakana UN, Marchetti E, Rappuoli R, Saul A, Martin LB, Necchi F, Podda A. Antibodies Elicited by the Shigella sonnei GMMA Vaccine in Adults Trigger Complement-Mediated Serum Bactericidal Activity: Results From a Phase 1 Dose Escalation Trial Followed by a Booster Extension. Front Immunol. 2021 May 4;12:671325. doi: 10.3389/fimmu.2021.671325. eCollection 2021. PMID 34017343
- [Derived] Launay O, Lewis DJM, Anemona A, Loulergue P, Leahy J, Scire AS, Maugard A, Marchetti E, Zancan S, Huo Z, Rondini S, Marhaba R, Finco O, Martin LB, Auerbach J, Cohen D, Saul A, Gerke C, Podda A. Safety Profile and Immunologic Responses of a Novel Vaccine Against Shigella sonnei Administered Intramuscularly, Intradermally and Intranasally: Results From Two Parallel Randomized Phase 1 Clinical Studies in Healthy Adult Volunteers in Europe. EBioMedicine. 2017 Aug;22:164-172. doi: 10.1016/j.ebiom.2017.07.013. Epub 2017 Jul 15. PMID 28735965
- [Derived] Muturi-Kioi V, Lewis D, Launay O, Leroux-Roels G, Anemona A, Loulergue P, Bodinham CL, Aerssens A, Groth N, Saul A, Podda A. Neutropenia as an Adverse Event following Vaccination: Results from Randomized Clinical Trials in Healthy Adults and Systematic Review. PLoS One. 2016 Aug 4;11(8):e0157385. doi: 10.1371/journal.pone.0157385. eCollection 2016. PMID 27490698

RESULTS

PARTICIPANT FLOW:
Groups:
- S. Sonnei 1790GAHB - 1 mcg: Subjects enrolled in COHORT A receiving 3 injections of S. sonnei 1790GAHB - 1 mcg
  S. sonnei 1790GAHB
- S. Sonnei 1790GAHB - 5 mcg: Subjects enrolled in COHORT B receiving 3 injections of S. sonnei 1790GAHB - 5 mcg
  S. sonnei 1790GAHB
- S. Sonnei 1790GAHB - 25 mcg: Subjects enrolled in COHORT C receiving 3 injections of S. sonnei 1790GAHB - 25 mcg
  S. sonnei 1790GAHB
- S. Sonnei 1790GAHB - 50 mcg: Subjects enrolled in COHORT D receiving 3 injections of S. sonnei 1790GAHB - 50 mcg
  S. sonnei 1790GAHB
- S. Sonnei 1790GAHB - 100 mcg: Subjects enrolled in COHORT E receiving 3 injections of S. sonnei 1790GAHB - 100 mcg
  S. sonnei 1790GAHB
- Placebo: 2 subjects enrolled in each COHORT A, B, C, D, E receiving 3 injections of Placebo. These were pooled in one Placebo group in the analyses
  Placebo
Period: Overall Study
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Started | 8 | 9 | 8 | 8 | 9 | 8
Completed | 8 | 9 | 8 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9 | 8 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 8 | 8 | 9 | 8 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (6.7) | 29.8 (7) | 26.8 (5.7) | 32.9 (7.7) | 26.9 (4.2) | 33.1 (8.2) | 30.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 4 | 4 | 7 | 28
  Male | 4 | 5 | 3 | 4 | 5 | 1 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 2 | 0 | 1 | 6
  White | 7 | 6 | 6 | 5 | 9 | 7 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 8 | 9 | 8 | 8 | 9 | 8 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Reaction After Any Vaccination
Description: Any erythema/induration refers to: ≥25 mm in diameter. Grade 3 (severe) refers to erythema/induration >100 mm in diameter. Grade 3 (severe) for injection site pain refers to: prevents daily activity
Time Frame: During a 7-day (Days 1-7) post vaccination period following any injection
Population: Analysis was done on as treated safety population
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9 | 8
Participants
  Any Pain | 8 | 9 | 8 | 8 | 9 | 6
  Grade 3 Pain | 0 | 0 | 0 | 1 | 1 | 0
  Any Erythema | 0 | 0 | 0 | 0 | 3 | 1
  Grade 3 Erythema | 0 | 0 | 0 | 0 | 1 | 0
  Any Induration | 0 | 0 | 0 | 2 | 2 | 0
  Grade 3 Induration | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited Systemic Reaction After Any Vaccination
Description: Any= Incidence of any symptom regardless of intensity grade. Grade 3 = symptom that prevented daily activities
Time Frame: During a 7-day (Days 1 to 7) post vaccination period following any injection
Population: Analysis was done on as treated population
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9 | 8
Participants
  Any Headache | 3 | 3 | 2 | 4 | 2 | 3
  Grade 3 Headache | 0 | 1 | 0 | 1 | 0 | 0
  Any Arthralgia | 2 | 0 | 2 | 3 | 3 | 1
  Grade 3 Arthralgia | 0 | 0 | 0 | 1 | 0 | 0
  Any Chills | 2 | 0 | 1 | 1 | 0 | 1
  Grade 3 Chills | 0 | 0 | 0 | 1 | 0 | 0
  Any Fatigue | 4 | 3 | 6 | 5 | 5 | 5
  Grade 3 Fatigue | 0 | 0 | 0 | 1 | 1 | 0
  Any Malaise | 0 | 1 | 0 | 1 | 2 | 0
  Grade 3 Malaise | 0 | 0 | 0 | 1 | 0 | 0
  Any Myalgia | 5 | 1 | 3 | 4 | 5 | 3
  Grade 3 Myalgia | 0 | 0 | 0 | 1 | 0 | 0
  Fever (≥38.0°C) | 1 | 0 | 0 | 0 | 0 | 0
  Fever (≥40.0°C) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Neutrophils Results Below and Above the Normal Ranges
Description: Day 8: VISIT 2 (D7 post 1st vac)
Time Frame: At Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9 | 8
Participants
  Neutrophils Results Below Normal Ranges | 0 | 1 | 0 | 1 | 0 | 0
  Neutrophils Results Above Normal Ranges | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Subjects With Neutrophils Results Below and Above the Normal
Description: Day 36: VISIT 3.1 (D7 post 2nd vac.)
Time Frame: At Day 36
Population: Some Arms have zero subjects attending visit 3.1, as complete blood counts testing 7 days after 2nd and 3rd vaccination was introduced following a protocol amendment while the study was ongoing.
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 5 | 8 | 3
Participants
  Neutrophils Results Below Normal Ranges | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Results Above Normal Ranges | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Subjects With Neutrophils Results Below and Above the Normal
Description: Day 57: VISIT 4 (3rd vac.)
Time Frame: At Day 57
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 7 | 8
Participants
  Neutrophils Results Below Normal Ranges | 0 | 1 | 0 | 1 | 0 | 0
  Neutrophils Results Above Normal Ranges | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Subjects With Neutrophils Results Below and Above the Normal
Description: Day 64: VISIT 4.1 (D7 post 3rd vac.)
Time Frame: At Day 64
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 2 | 7 | 4
Participants
  Neutrophils Results Below Normal Ranges | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Results Above Normal Ranges | 0 | 0 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Subjects With Neutrophils Results Below and Above the Normal
Description: Day 85: VISIT 5 (1 month post 3rd vac.)
Time Frame: At Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 6 | 8 | 8
Participants
  Neutrophils Results Below Normal Ranges | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils Results Above Normal Ranges | 0 | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Number of Subjects With Neutrophils Results Below and Above the Normal
Description: Day 225: VISIT 6 (6 months post 3rd vac.)
Time Frame: At Day 225
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 8 | 8
Participants
  Neutrophils Results Below Normal Ranges | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils Results Above Normal Ranges | 0 | 0 | 1 | 0 | 1 | 1

9. Secondary Outcome: Anti-LPS S. Sonnei Serum IgG Geometric Mean Concentration (GMCs)
Time Frame: At baseline, at 28 days after each vaccination and at 168 days after last vaccination
Population: Analysis was done on the Full Analysis Set (FAS), ie, subjects in All Enrolled Set who: received a study vaccination, provided evaluable serum, with results available & who was not excluded due to protocol deviations or other reasons defined before unblinding or analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 9 | 8
Titers
  Baseline (Day 1) | 4.71 [2.02 to 11] | 7.74 [2.72 to 22] | 27 [3.75 to 191] | 8.78 [1.2 to 64] | 6.91 [2.03 to 24] | 6.37 [2.38 to 17]
  One month after first vac. | 6.2 [1.97 to 20] | 23 [6.13 to 86] | 141 [21 to 962] | 186 [40 to 855] | 157 [45 to 546] | 6.35 [2.61 to 15]
  One month after second vac.: number analyzed (Participants) | 8 | 9 | 8 | 6 | 8 | 8
  One month after second vac. | 18 [6.95 to 49] | 41 [11 to 148] | 314 [60 to 1646] | 111 [17 to 717] | 193 [52 to 707] | 6.56 [2.5 to 17]
  One month after third vac.: number analyzed (Participants) | 8 | 9 | 7 | 6 | 8 | 8
  One month after third vac. | 32 [10 to 98] | 67 [17 to 269] | 486 [120 to 1959] | 149 [17 to 1289] | 159 [47 to 539] | 7.71 [2.31 to 26]
  Six months after third vac.: number analyzed (Participants) | 8 | 9 | 7 | 6 | 8 | 7
  Six months after third vac. | 12 [2.66 to 57] | 42 [9.96 to 178] | 418 [87 to 2002] | 106 [9.89 to 1143] | 102 [27 to 383] | 5.05 [1.65 to 15]

10. Secondary Outcome: Number of Subjects With Seroresponse for Anti-LPS S. Sonnei
Description: Seroresponse is defined as: If half of the baseline value is greater than 25 ELISA Unit (EU) then an increase of at least 50% in the post-vaccination sample as compared to baseline [i.e. ((Post-vac minus baseline)/baseline)100% ≥ 50%]. If half of the baseline value is less or equal to 25 EU then an increase of at least 25 EU in the post-vaccination sample as compared to baseline (i.e. [post-vac minus baseline] ≥25 EU)
Time Frame: At 28 days after each vaccination and 168 days after last vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 9 | 8
Participants
  One month after first vac. | 1 | 3 | 5 | 6 | 8 | 0
  One month after second vac.: number analyzed (Participants) | 8 | 9 | 8 | 6 | 8 | 8
  One month after second vac. | 2 | 5 | 7 | 4 | 7 | 0
  One month after third vac.: number analyzed (Participants) | 8 | 9 | 7 | 6 | 8 | 8
  One month after third vac. | 3 | 7 | 6 | 4 | 7 | 1
  Six months after third vac.: number analyzed (Participants) | 8 | 9 | 7 | 6 | 8 | 7
  Six months after third vac. | 2 | 6 | 6 | 4 | 6 | 0

11. Secondary Outcome: Number of Subjects With High Seroresponse for Anti-LPS S. Sonnei (IgG ELISA ≥121 EU)
Description: High seroresponse is defined as a post vaccination titer ≥X anti-LPS serum IgG units in the GSK (former Novartis) ELISA that correspond to a titer of 1:800 in the ELISA method used by Cohen et al. To determine the value for 'X' the GSK (former Novartis) anti-LPS ELISA was calibrated against the Cohen ELISA and it was found that a concentration of 121 EU EU/mL corresponds to a titer of 1:800 in the Cohen assay
Time Frame: At baseline, at 28 days after each vaccination and at 168 days after last vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 9 | 8
Participants
  Baseline | 0 | 0 | 2 | 2 | 1 | 0
  One month after first vac. | 0 | 2 | 6 | 4 | 4 | 0
  One month after second vac.: number analyzed (Participants) | 8 | 9 | 8 | 6 | 8 | 8
  One month after second vac. | 1 | 3 | 6 | 3 | 5 | 0
  One month after third vac.: number analyzed (Participants) | 8 | 9 | 7 | 6 | 8 | 8
  One month after third vac. | 2 | 5 | 6 | 4 | 4 | 0
  Six months after third vac.: number analyzed (Participants) | 8 | 9 | 7 | 6 | 8 | 7
  Six months after third vac. | 2 | 2 | 5 | 3 | 3 | 0

ADVERSE EVENTS:
Time Frame: Solicited reactions were reported in 7-day post vaccination period (i.e. Day 1 to Day 7, Day 29 to Day 35, and Day 57 to Day 63). Unsolicited Adverse Events were reported during a 28-day post vaccination period (i.e. Day 1 to Day 28, Day 29 to Day 56, and Day 57 to Day 84). AEs leading to study withdrawal, SAEs and AEs of special interest (reactive arthritis) were reported during all study period (i.e. Day 1 to Day 225).
Arm/Group | S. Sonnei 1790GAHB - 1 mcg | S. Sonnei 1790GAHB - 5 mcg | S. Sonnei 1790GAHB - 25 mcg | S. Sonnei 1790GAHB - 50 mcg | S. Sonnei 1790GAHB - 100 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8 | 8/8 | 9/9 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S. Sonnei 1790GAHB - 1 mcg (N=8) | S. Sonnei 1790GAHB - 5 mcg (N=9) | S. Sonnei 1790GAHB - 25 mcg (N=8) | S. Sonnei 1790GAHB - 50 mcg (N=8) | S. Sonnei 1790GAHB - 100 mcg (N=9) | Placebo (N=8)
Rhinoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (6) | 3 (8) | 6 (8) | 5 (13) | 5 (9) | 5 (11)
Injection site erythema (General disorders) | 3 (6) | 0 (0) | 3 (6) | 5 (9) | 7 (14) | 2 (2)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (7) | 6 (12) | 2 (4)
Injection site pain (General disorders) | 8 (20) | 9 (19) | 8 (23) | 8 (22) | 9 (26) | 6 (17)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (13) | 3 (13) | 5 (7) | 5 (12) | 2 (3) | 5 (14)
Morton's neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 2 (3) | 3 (5) | 3 (6) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (5) | 4 (7) | 5 (10) | 3 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

Trial results may not be published or disclosed in any other way by the Institution, without the prior written consent by the Sponsor.